CLINICAL TRIAL: NCT06546605
Title: Evaluating the Effects of Diverse Training Methods on Athletic Performance and Health: A Randomized Crossover Study
Brief Title: A Randomized Crossover Study on Diverse Training Methods to Enhance University Athletes' Performance and Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Macau (Other)
Responsible Party: Principal Investigator, Siman Lei, Assistant Professor, University of Macau
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HE-0151-2024
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-10

CONDITIONS: Athletic Performance; Plyometric Exercise; Healthy
Keywords: Plyometric Training; Functional Training; Whole-Body Electrical Muscle Stimulation (WB-EMS); Injury Prevention; Randomized Crossover Study; Athletic Performance; Functional Movement Skills
MeSH Terms: interventions — Emergency Treatment; Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Plyometric Training to WB-EMS Training Group (PTG-ETG) (Experimental): Participants in the PTG-ETG will undergo a progressive plyometric training program in the first 8-week intervention period, followed by a WB-EMS training program in the second 8-week intervention period after the crossover. The plyometric training will include exercises such as box jumps, depth jumps, split squat jumps, and single-leg hops to enhance lower extremity power, speed, and agility.
  After the crossover, participants will engage in a WB-EMS training program that combines dynamic exercises with concurrent electrical stimulation using the miha bodytec® device. Each WB-EMS session will consist of a warm-up followed by 4-6 exercises lasting 4-6 seconds each, with 4 seconds of rest between exercises. The intensity of the electrical stimulation will be set at 70-85% of the participant's maximal comfort level and adjusted based on individual tolerance. The WB-EMS training will be performed twice a week for 20-25 minutes per session during the second intervention period.
  Interventions: Device: Whole-Body Electrical Muscle Stimulation (WB-EMS) Training; Behavioral: Plyometric Training
- Functional Training to Plyometric Training Group (FTG-PTG) (Experimental): Participants in the FTG-PTG will engage in a functional training program tailored to their specific sport in the first 8-week intervention period, followed by a progressive plyometric training program in the second 8-week intervention period after the crossover. The functional training will incorporate sport-specific movements, such as multidirectional lunges, rotational medicine ball throws, and single-leg balance drills.
  After the crossover, participants will undergo a progressive plyometric training program designed to enhance their lower extremity power, speed, and agility. The program will include a variety of plyometric exercises such as box jumps, depth jumps, split squat jumps, and single-leg hops.
  Each session will begin with a dynamic warm-up, then proceed to the main exercise, and then cool down with stretching.
  Interventions: Behavioral: Plyometric Training; Behavioral: Functional Training
- WB-EMS Training to Functional Training Group (ETG-FTG) (Experimental): Participants in the ETG will participate in a training program that combines dynamic exercises with concurrent WB-EMS. The WB-EMS device (miha bodytec®, Augsburg, Germany) will be used to apply electrical stimulation to major muscle groups while participants perform exercises such as squats, lunges, and trunk rotations. Each session will consist of a warm-up followed by 4-6 WB-EMS exercises lasting 4-6 seconds each, with 4 seconds of rest between exercises. The intensity of the electrical stimulation will be set at 70-85% of the participant's maximal comfort level and adjusted based on individual tolerance. The WB-EMS training will be performed twice a week for 20-25 minutes per session.
  After the crossover, participants will engage in a functional training program that simulates game-specific movements, such as multidirectional lunges, rotational medicine ball throws, and single-leg balance drills.The program will also include core stability and injury prevention exercises.
  Interventions: Device: Whole-Body Electrical Muscle Stimulation (WB-EMS) Training; Behavioral: Functional Training
- Control Group (CG) (No Intervention): Participants in the CG will maintain their usual team training routines and practices throughout the study period, without receiving any additional training interventions. They will serve as a reference to compare the effects of the plyometric, functional, and WB-EMS training programs on athletic performance and health-related outcomes. Participants in this group will undergo all scheduled assessments at baseline, after each 8-week intervention period, and during the follow-up to track changes in their performance and health status over time. The control group will help determine the extent to which changes in the intervention groups can be attributed to the specific training programs, rather than other factors such as natural progression or regular team training.

INTERVENTIONS:
Device: Whole-Body Electrical Muscle Stimulation (WB-EMS) Training — Whole-Body Electrical Muscle Stimulation (WB-EMS) Training is a novel training modality that involves the simultaneous electrical stimulation of multiple muscle groups while performing dynamic exercises. Participants in the WB-EMS Training Group will use the miha bodytec device (Augsburg, Germany), which consists of a special suit with integrated electrodes covering major muscle groups. The device generates electrical impulses (85 Hz, 350 μs) that cause involuntary muscle contractions during exercises like squats, lunges, and trunk rotations.Each 20-25-minute WB-EMS session will be conducted twice a week during the two 8-week intervention periods. Sessions will include a warm-up followed by 4-6 WB-EMS exercises performed for 4-6 seconds each, with 4 seconds of rest between exercises. The intensity of the stimulation and exercises will be progressively increased based on individual adaptation and tolerance, with the stimulation intensity set at 70-85% of the maximal tolerable level.
  Other Names: Electrical Myostimulation (EMS) Training; Neuromuscular Electrical Stimulation (NMES) Training; Full-Body Electromyostimulation Training
  Arms: Plyometric Training to WB-EMS Training Group (PTG-ETG); WB-EMS Training to Functional Training Group (ETG-FTG)
Behavioral: Plyometric Training — Plyometric Training is a high-intensity, explosive strength training modality that involves quick, powerful movements designed to increase muscle power, speed, and agility. Participants in the Plyometric Training Group will engage in a progressive plyometric training program that emphasizes eccentric muscle loading followed by rapid concentric contractions.
  The plyometric exercises will include various types of jumps, hops, and bounds, such as box jumps, depth jumps, split squat jumps, and single-leg hops. Each training session will begin with a dynamic warm-up, followed by 4-6 plyometric drills performed for 3-5 sets of 8-12 repetitions, with 60-90 seconds of rest between sets. The intensity and volume of the exercises will be gradually increased over the two 8-week intervention periods.
  Other Names: Reactive Strength Training; Stretch-Shortening Cycle Training
  Arms: Functional Training to Plyometric Training Group (FTG-PTG); Plyometric Training to WB-EMS Training Group (PTG-ETG)
Behavioral: Functional Training — Functional Training is a training approach that focuses on exercises that simulate the demands of specific sports or daily activities, targeting multiple muscle groups and movement patterns simultaneously. Participants in the Functional Training Group will engage in a tailored functional training program designed to enhance their performance in basketball or volleyball.
  The functional training exercises will incorporate multi-joint, multi-planar movements that mimic game-specific actions, such as multidirectional lunges, rotational medicine ball throws, and single-leg balance drills. Each session will start with a dynamic warm-up, followed by 6-8 functional exercises performed for 3-4 sets of 8-12 repetitions, with 60 seconds of rest between sets. The program will also include core stability and injury prevention exercises.
  Other Names: Movement-Based Training; Sport-Specific Training
  Arms: Functional Training to Plyometric Training Group (FTG-PTG); WB-EMS Training to Functional Training Group (ETG-FTG)

SUMMARY:
The goal of this randomized crossover study is to investigate the effects of plyometric training, functional training, and whole-body electrical muscle stimulation (WB-EMS) on athletic performance and health in university basketball and volleyball players. The main questions it aims to answer are:

1. Which training modality (plyometric, functional, or WB-EMS) leads to the greatest improvements in athletic performance measures such as power, speed, and agility?
2. How do these training modalities compare in terms of their effects on overall health, injury risk reduction, and psychological well-being?

Researchers will use a crossover design, where each participant experiences multiple training modalities in a sequential manner, to provide a more rigorous and comprehensive evaluation of the interventions' effectiveness.

Participants will:

1. Be randomly assigned to one of four training sequences, each consisting of two 8-week intervention periods separated by a 4-week washout phase;
2. Experience at least two of the three training modalities (plyometric, functional, or WB-EMS) during the intervention periods;
3. Maintain their regular training routines if assigned to the control group;
4. Undergo assessments, including anthropometric measurements, physical fitness tests, and questionnaires, at baseline, after each intervention period, and during a follow-up session.

The findings of this study will provide valuable insights into the optimal sequencing and combination of training modalities to maximize athletic performance and promote health among university basketball and volleyball players.

DETAILED DESCRIPTION:
Background: Enhancing athletic performance and reducing injury risk require effective training techniques. University athletes, often practicing only 2-3 times a week, need support to reach optimal fitness. This study examines the effects of plyometric, functional, and WB-EMS training on the health and performance of collegiate basketball and volleyball players.

Objective: The primary aim is to evaluate the effectiveness of these training modalities in improving athletic performance metrics such as strength, speed, agility, and endurance. Secondary aims include determining their influence on recovery and injury prevention and exploring potential differences in response among athletes from different sports disciplines.

Study Design: This is a randomized crossover study. Participants will be randomly allocated to one of four groups: plyometric training, WB-EMS training, functional training, or control group. The intervention will consist of two 8-week training periods separated by a 4-week washout period.

Participants: 120 male and female basketball and volleyball players aged 18-30 from University teams in Macau will be recruited. They should have at least 3-4 years of competitive experience in their respective sports.

Interventions: The plyometric group will focus on explosive movements and jumps. The WB-EMS group will perform exercises while receiving electrical stimulation. The functional training group will engage in sport-specific exercises. The control group will maintain their regular training. Each session will include a warm-up, specific exercises, and a cool-down.

Outcome Measures: Participants will undergo assessments at baseline, post-intervention, and follow-up. These include anthropometric measurements, physical fitness tests (e.g., Y-Balance Test, FMS, 1RM half-squat, leg muscle volume, vertical jump, agility, sprint), and questionnaires (e.g., ERQ, PSQI, SES, SWLS).

Statistical Analysis: Mixed-design ANOVA or ANCOVA will compare the effects across time points. Post-hoc tests will determine specific differences between groups and time points. Significance will be set at p value smaller than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Team Membership: Participants must be officially registered members of the Macau universities' 's men's and women's basketball or volleyball teams.
2. Age Range: Participants must be aged between 18 and 30 years.
3. Health Status: Participants should be in good health, free from any chronic diseases, serious health conditions, or contraindications that could impair their athletic performance, preclude their safe participation in the study, or present undue risks when exposed to WB-EMS. Participants must provide informed consent and be willing to undergo WB-EMS training after being fully apprised of the potential risks and benefits.
4. Commitment: Participants must be able to engage fully in the intervention period and all associated assessments.
5. Experience: Participants are required to have a minimum of three to four years of competitive basketball or volleyball experience.

Exclusion Criteria:

1. Unable to provide informed consent.
2. Unwillingness to be allocated to one of the four groups.
3. Have suffered a lower extremity injury or required surgery within the past 6 months.
4. Have undergone electrical stimulation training for the previous six months.
5. Have been diagnosed with a cardiovascular or neurological disease or abnormality.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-10-03 (Estimated)

PRIMARY OUTCOMES:
Squat Jump (SJ) Test | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The squat jump is a performance test used to measure the explosive power of an athlete's lower extremities, particularly focusing on the ability to generate force from a static position. Participants begin by standing with their feet shoulder-width apart, then descend into a squat position until their thighs are parallel to the ground. From this static squat position, they explosively jump as high as possible without the assistance of arm movement. This test typically involves performing two jumps, with a 45-second rest interval between jumps. The highest jump (cm) from the two attempts is recorded. A three-dimensional force platform, the Just Jump system NO101 (Probotics Inc.), is commonly used to measure and collect height data during the jumping process. The test is significantly correlated with explosive power and athletic performance, demonstrating excellent reliability with an intra-session ICC of 0.97 and an inter-session ICC of 0.94.
Countermovement Jump（CMJ） | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  Participants are required to stand with their feet shoulder-width apart, toes slightly pointing outwards, and hands placed on their hips to prevent arm movement, allowing for an accurate assessment of lower extremity explosive power. At the start of the test, participants rapidly bend their knees, lowering their center of gravity until their knees reach approximately a 90-degree angle, then quickly extend their knee, hip, and ankle joints, jumping upwards with maximum effort. Each movement is performed twice, with a 45-second rest interval between jumps. The best jump height data (cm) is recorded. Jump height data during the jumping process is collected using a three-dimensional force platform NO101 (Just Jump, Probotics Inc.). The CMJ is a widely used and validated method for assessing jumping ability and explosive power, demonstrating good reliability and validity with an intra-session ICC of 0.95 and an inter-session ICC of 0.93.
Running Jump Off Test | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The running jump off test requires participants to first stand directly beneath the apparatus, with their feet flat on the ground and one arm extended upwards to measure their standing reach height. The subject then stands approximately 15 feet (about 5 meters) from the base of the apparatus. In preparation for the jump, they take 3 to 5 steps, then take off from both legs (or a single leg, depending on the specific requirements of the test), using their arms to help propel their body upwards. The goal is to have the body positioned directly beneath the apparatus at the peak of the jump, with arms fully extended, which may require some practice to perfect the timing and takeoff point. The difference between the standing reach height and the highest point touched during the jump is recorded, with the best result (cm) from three attempts being noted. The vertical jump apparatus is used, demonstrating good reliability with an ICC ranging from 0.90 to 0.96.
Modified 505 Change of Direction Test | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The 505 Change of Direction (COD) test, performed from a stationary start, evaluates an athlete's ability to execute a rapid 180° turn within a 5-meter distance. The athlete begins the test from a standing position, placing their preferred foot half a meter behind the starting line and using this foot as the turning pivot. Each athlete performs three attempts, with the fastest completion time (s) recorded using precise timing equipment. A two-minute rest period is provided between each trial. According to the definition by Nimphius et al., the change of direction deficit (CODDEF) for the 505 test is determined using the following formula: CODDEF = (Modified 505 test time - 10-meter sprint time). This test demonstrates good reliability with an ICC of 0.87 and is highly correlated with the standard 505 test, with a correlation coefficient (r) of 0.87.
Sprint 4 × 5 m Test | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The setup requires 5 cones placed 5m apart. The subject stands with feet apart, straddling a cone between their legs. Upon hearing an auditory signal, they run 5 meters to point A; then turn 90° to the right and run 5 meters to point B. After the second 90° turn, they run to point C, where they make a 180° turn and run to the finish line. Each athlete performs three attempts, with the fastest completion time (s) recorded using precise timing equipment. A two-minute rest period is provided between each trial. This test demonstrates good reliability with an ICC ranging from 0.88 to 0.91.
Modified Agility T-Test (MAT) | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The Modified Agility T-Test (MAT), developed by Radhouane et al., is based on the traditional T-test and aims to assess an athlete's ability to quickly change direction, including forward sprinting, lateral shuffling, and backward movement. MAT adjusts the spatial layout of the original T-test, reducing the total running distance from 36.56 meters to 20 meters while maintaining the same types of movements and number of direction changes, adapting to space-constrained environments. Each athlete performs three attempts, with the fastest completion time (s) recorded using precise timing equipment. A two-minute rest period is provided between each trial. The test has high reliability with an ICC ranging from 0.82 to 0.96 and is highly correlated with the standard T-test, with a correlation coefficient (r) of 0.92, effectively differentiating athletes' agility performance.

SECONDARY OUTCOMES:
Functional Movement Screening (FMS) | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The FMS Functional Movement Screening Test Tool (FMS, Perform Better, USA) is a system that assesses an individual's motor control stability, body balance, flexibility, and proprioception when completing basic movement patterns. As shown in Table 3, the following is a brief operation process and scoring standard for the seven basic movements of the FMS test. Each item is scored from 0 to 3 points, with a total score of 0 to 21 points. 0 points: Pain occurs during the test; 1 point: Unable to complete. The movement may not be able to maintain the starting posture; 2 points: Able to complete the movement, but the quality of the movement is not high; 3 points: The movement is completed with high quality. Functional movement screening is completed using the FMS test kit. The FMS is a widely used and validated method for measuring human dynamic balance and assessing injuries, demonstrating good reliability and validity with an ICC ranging from 0.87 to 0.98.
Y balance test (YBT) | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The subjects stood barefoot on one leg using a test instrument (Y-balance, Performance Health, USA). The non-supporting leg was stably extended to the farthest distance in three directions: forward, backward inward, and backward outward, and held for 3 seconds. Practice 3 times on each side before the test, rest for 5 minutes before officially starting the test, and test 3 times in each direction. The test index is the relative value of the legs on each side. Relative value of each leg (%) = (anterior + posteromedial + posterolateral) / (3*leg length in lateral lying position). The higher the relative value of each leg means better lower limb dynamic balance ability, and more Optimum lower limb mobility and flexibility, and potentially lower risk of lower limb injury.The Y balance test is a widely used and validated method for measuring human dynamic balance and assessing injuries, demonstrating good reliability and validity with an ICC ranging from 0.91 to 0.99.
Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report measure of sleep quality, containing 18 self-rated items across seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is scored on a scale of 0-3, with a total score range of 0-21 for the seven components. Higher scores indicate poorer sleep quality. The scale has demonstrated good internal consistency reliability, with a Cronbach's α ranging from 0.80 to 0.83, and a test-retest reliability ranging from 0.85 to 0.87. Liu Xianchen et al. conducted a Chinese revision and validation of the PSQI, confirming that the Chinese version is an effective tool for assessing sleep quality.
Self-Efficacy Scale (SES) | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The Self-Efficacy Scale (SES) is a 13-item self-report scale designed to assess an individual's beliefs about their own capabilities. Each item is scored on a scale ranging from 1 (strongly disagree) to 7 (strongly agree), with a total score range of 13-91 for the 13 items. Higher scores indicate stronger self-efficacy. The scale has an internal consistency reliability (Cronbach's α) of 0.91. The SES was originally developed by Schwarzer and Jerusalem and has been widely applied across different cultural contexts.
Satisfaction With Life Scale (SWLS) | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8weeks for phase 2）
  The Satisfaction With Life Scale (SWLS) is a brief 5-item self-report scale used to assess an individual's overall satisfaction with their life. Each item is scored on a scale ranging from 1 (strongly disagree) to 7 (strongly agree), with a total score range of 5-35 for the 5 items. Higher scores indicate greater life satisfaction. The SWLS has an internal consistency reliability (Cronbach's α) of 0.87 and is positively correlated with multiple indicators of well-being, supporting its validity. Wu Minglong conducted a Chinese revision and cross-cultural validation of the SWLS, and the results demonstrated that the Chinese version of the SWLS also has good reliability and validity.
Emotion Regulation Questionnaire (ERQ) | From enrollment to the end of intervention at 20 weeks（8 weeks for phase 1,4 weeks for wash out and 8 weeks for phase 2）
  The Emotion Regulation Questionnaire (ERQ) is a 10-item self-report scale used to assess an individual's habitual use of two emotion regulation strategies: expressive suppression and cognitive reappraisal. Each item is scored on a scale ranging from 1 (strongly disagree) to 7 (strongly agree), with a total score range of 10-70 for the 10 items. Higher scores indicate a greater tendency to use the corresponding emotion regulation strategy. The scale contains two subscales: expressive suppression (4 items) and cognitive reappraisal (6 items). The internal consistency reliability for these subscales is strong, with Cronbach's α values ranging from 0.73 to 0.79 for expressive suppression and from 0.75 to 0.82 for cognitive reappraisal. Wang Dandan et al. conducted a Chinese revision of the ERQ, also demonstrated good psychometric properties. In this study, the questionnaire is primarily distributed to subjects in paper form, to be completed within one hour after testing and training.

CONTACTS AND LOCATIONS:
Locations (2):
- Macau (2):
  - UM Sports Complex (N8) , Avenida da Universidade Taipa, Macau, China, Macao
  - University of Macau, Taipa

IPD SHARING:
Plan to Share IPD: No